CLINICAL TRIAL: NCT05362812
Title: Prediction of Lupus Renal Flares Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Enghard, PD Dr. med, Charite University, Berlin, Germany
Other Study IDs: PreLuFlare
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Lupus Nephritis; Flow Cytometry; CD4-Positive T-Lymphocytes; Biomarker; Urine Specimen Collection
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, lymphocytes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with systemic lupus erythematosus: Diagnostic Test: Flow cytometry analysis of urine samples. Urine samples will be conserved and frozen upon arrival. All samples will be stained according to T cell and B cell panel with fluorochromes. T cell panel: CD3, CD4, CD8, CCR7, CD45RO, CD38, CD279; B cell panel: CD19, CD20, CD27, CD38, CD21, IgD, CXCR5

SUMMARY:
In patients with systemic lupus erythematosus, urinary CD4+ T cells may have the potential to predict subsequent renal flares in the next 6 months. Patients with systemic lupus erythematosus from our outpatient clinic will be included in this cross-sectional, prospective biomarker study regardless of disease activity, clinical phenotype, and disease duration or baseline therapy. Urinary T cells will be analyzed by flow cytometry. 6 months after sample collection a clinical follow-up will be conducted to assess the occurrence of either recurrent or de novo renal flares.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosis of SLE according to the 2019 EULAR/ACR classification criteria Stable immunosuppressive or biologic background therapy within the last 6 months prior to inclusion

Exclusion Criteria:

* Age < 18
* Inability to consent
* Urinary tract infection (defined by detection of nitrite or positive urine culture)
* Patients on chronic dialysis
* Concomitant other autoimmune disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus from the outpatient clinic of the Department of Rheumatology and Clinical Immunology, University Hospital Charité, Berlin
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Renal flares within the next 6 months | 6 months
  To evaluate whether the number of urinary CD4+ T cells has the potential to predict subsequent renal flares in the next 6 months.
  Renal flares will be defined as an increase of proteinuria by > 0.5 g/g creatinine or an increase in creatinine by 30% without other likely explanation or a novel kidney biopsy demonstrating lupus nephritis.

SECONDARY OUTCOMES:
To investigate whether the phenotype of urinary T cell subsets can predict renal involvement or subsequent renal flares in preexisting LN (CD4+ and CD8+ T cells subsets). | 6 months
To investigate whether the number and phenotype of urinary B- and plasma cell subsets can predict renal involvement or subsequent renal flares in preexisting LN | 6 months
To evaluate whether increased surface expression of CD38 on peripheral blood memory T cells is associated with the presence of renal involvement. | 6 months
To assess whether urinary or peripheral blood T- and B cell subsets or IFN-I activity can predict the incidence of mild/moderate or severe flares of SLE according to the SELENA-SLEDAI Flare Index (SFI) | 6 months
Investigate whether Belimumab treatment has a beneficial impact on biomarkers associated with renal flares and loss of renal function. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Enghard, MD, Principal Investigator — Department of Nephrology and Intensive Care, Charite University Hospital; Tobias Alexander, MD, Principal Investigator — Department of Rheumatology and Clinical Immunology, Charite University Hospital
Locations (1):
- Department of Nephrology and Intensive Care, Charite University Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Enghard P, Rieder C, Kopetschke K, Klocke JR, Undeutsch R, Biesen R, Dragun D, Gollasch M, Schneider U, Aupperle K, Humrich JY, Hiepe F, Backhaus M, Radbruch AH, Burmester GR, Riemekasten G. Urinary CD4 T cells identify SLE patients with proliferative lupus nephritis and can be used to monitor treatment response. Ann Rheum Dis. 2014 Jan;73(1):277-83. doi: 10.1136/annrheumdis-2012-202784. Epub 2013 Mar 8. PMID 23475982
- [Background] Rose T, Grutzkau A, Klotsche J, Enghard P, Flechsig A, Keller J, Riemekasten G, Radbruch A, Burmester GR, Dorner T, Hiepe F, Biesen R. Are interferon-related biomarkers advantageous for monitoring disease activity in systemic lupus erythematosus? A longitudinal benchmark study. Rheumatology (Oxford). 2017 Sep 1;56(9):1618-1626. doi: 10.1093/rheumatology/kex220. PMID 28859328
- [Background] Burns M, Ostendorf L, Biesen R, Grutzkau A, Hiepe F, Mei HE, Alexander T. Dysregulated CD38 Expression on Peripheral Blood Immune Cell Subsets in SLE. Int J Mol Sci. 2021 Feb 28;22(5):2424. doi: 10.3390/ijms22052424. PMID 33670902